CLINICAL TRIAL: NCT06000943
Title: Ischemic And Bleeding Risk Assessment After TAVR (FOCUS ONE Registry)
Brief Title: Ischemic And Bleeding Risk Assessment After TAVR
Acronym: FOCUS ONE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Niguarda Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: F1R
Record Dates: First submitted 2023-08-02; First posted 2023-08-21 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Aortic Valve Stenosis; Transcatheter Aortic Valve Replacement
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Lower Surgical Risk: Surgical risk stratification. All the following groups will be define according with STS and Euroscore II score and stratified based on antithrombotic strategy in all possible combinations (SAPT, DAPT, OAC, OAC+SAPT)
  Interventions: Other: Low vs Intermediate vs High surgical risk stratified according with SAPT/DAPT/OAC and OAC+SAPT
- Intermediate Surgical Risk: Surgical risk stratification. All the following groups will be define according with STS and Euroscore II score and stratified based on antithrombotic strategy in all possible combinations (SAPT, DAPT, OAC, OAC+SAPT)
  Interventions: Other: Low vs Intermediate vs High surgical risk stratified according with SAPT/DAPT/OAC and OAC+SAPT
- High Surgical Risk: Surgical risk stratification. All the following groups will be define according with STS and Euroscore II score and stratified based on antithrombotic strategy in all possible combinations (SAPT, DAPT, OAC, OAC+SAPT)
  Interventions: Other: Low vs Intermediate vs High surgical risk stratified according with SAPT/DAPT/OAC and OAC+SAPT

INTERVENTIONS:
Other: Low vs Intermediate vs High surgical risk stratified according with SAPT/DAPT/OAC and OAC+SAPT — All patients undergoing TAVR will be stratified according with surgical risk level and all combination of antithrombotic therapy at discharge
  Low risk (SAPT vs DAPT and OAC vs OAC+SAPT) Intermediate risk (SAPT vs DAPT and OAC vs OAC+SAPT) High risk (SAPT vs DAPT and OAC vs OAC+SAPT)

SUMMARY:
Transcatheter aortic valve replacement (TAVR) represents an effective treatment to improve symptoms and prognosis in patients with symptomatic severe aortic stenosis (AS) (1-2).

Giving an established uniform approach towards anticoagulation and antithrombotic therapy after TAVR in the post POPULAR-TAVI era, recent data coming from the analysis of different trials, highlight the relevance of the patient's background on the occurrence of ischemic and bleeding events.

Despite this a targeted antithrombotic strategy remains unexplored and all patients undergoing TAVR without other indication to DAPT or OAC, were currently treated according with the concept of "less is more" (only SAPT or only OAC) regardless the risk level (5-6).

The keys points of the project will be 1) the assessment of ischemic and bleeding risk after TAVR stratified according with antithrombotic therapy and surgical risk; 2) the evaluation of the impact of prostheses type and the complete blood count variables (hemoglobine and platelets) on the daily average ischemic and bleeding risk and 3) the evaluation of the dynamic therapeutic changes after TAVR during the follow up.

DETAILED DESCRIPTION:
Nowadays in the post POPULAR-TAVI era, after transcatheter aortic valve replacement (TAVR), an establish uniform approach towards anticoagulation and antithrombotic therapy were established.

All patients undergoing TAVR without other indication to dual antiplatelet therapy (DAPT) or oral anticoagulation (OAC), were currently treated according with the general concept of "less is more" (only single antiplatelet therapy - SAPT or only oral anticoagulation - OAC) [1-3].

By comparing the frequency of ischemic and bleeding events, data from trial revealed that the bleeding events were more frequent than the ischemic one despite the level of surgical risk, however a gradient of reduction in terms of difference was seen from the highest to the lowest risk profile [4].

Furthermore, recent literature showed how the timeframe analysis approach, giving the possibility for a complete time variability evaluation, is able to visualize the fluctuation of the risk over the time. Unfortunately, no stratified data according with the surgical risk level, are available using this approach [5].

Moreover, despite these results that highlight the relevance of the patient's background on the occurrence of ischemic and bleeding events, a tailored antithrombotic strategy remains unexplored and all patients undergoing TAVR without other indication to DAPT or OAC, were currently treated with a uniform approach in terms of intensity during the time (1-3).

1.1. Assessment of ischemic and bleeding risk after TAVR according with antithrombotic therapy and surgical risk The rate of adverse thrombotic and hemorrhagic events occurred in the first days after the procedure, were mainly driven by the TAVR's access bleeding and the periprocedural stroke.

Recent study, using the average daily risk analysis, showed the prevalence of the ischemic risk in the first 30 days after the procedure followed by a rising of the bleeding one which become predominant during the follow up, affecting the long-term prognosis [5].

However, only data based on surgical risk derived from the 'first time event approach' are available in the literature and none of them investigates whether the higher expected risks - both ischemic and hemorrhagic - in the highest risk cohort remain high even months after TAVR.

Bearing this in mind, these observations revealed that ischemic and bleeding events are not evenly distributed over time, suggesting that a risk-based modulation of the antithrombotic therapy could be better capture the time-dependent evolution of the phenomena. Experience from several studies on antithrombotic therapy in the PCI field, have focused on the intensity and the timing of administration, while no such evidence exists in the field of TAVR (6-7).

Thus, the comprehension of this phenomena holds the potential benefit of a tailored antithrombotic therapy guided by an integrated approach based on the trend of ischemic and bleeding risk stratified according to the patient's risk profile and the antithrombotic regimen adopted.

1.2. Impact of prostheses type and complete blood count variables on ischemic and bleeding events As the same of patient's features and periprocedural variables, it is possible to assume that also the prostheses characteristics in terms of type of leaflet (porcine vs bovine), stent frame amount (short frame versus long frame) and the number of they (valve-in-valve), are not fully investigated previously and may play a role in the thrombotic and hemorrhagic adverse events occurrence.

Understanding the impact of structural and functional valve's characteristics on the bleeding and ischemic risk among patients who undergo TAVR, may have important implications in prosthesis and antithrombotic therapy selection and needs to be investigated properly with a "repeated-event" analysis.

Moreover, also the frequent phenomenon of anemia and thrombocytopenia after TAVR, were identified from several studies as predictors of poor outcome up to 1 year follow up even with a perfect prosthesis function and despite the mechanism behind, it's not completely understood (8). According to these data the relationship between blood count abnormalities, type of prosthesis and ischemic and bleeding risk have never been explored.

The identification of predictive variables leading to the development of anemia and thrombocytopenia and their impact on the risk of hemorrhagic and thrombotic events, might allow us a tailored selection of prosthesis, antithrombotic strategy and procedural planning in order to potentially reduce the risk of adverse events.

1.3. Dynamic therapeutic changes after TAVI Several studies investigated the impact of different antithrombotic strategies on outcomes and prosthesis performance by comparing different approaches in combination. However, most of them assessed the clinical endpoints considering only the discharge therapy, with a lack of real data in terms of regimes switching and duration of any effective treatment prescribed.

The assessment of these data during follow-up, remains underexplored even though their availability could potentially allow an accurate definition of the ongoing strategy at the time of adverse event occurrence. Moreover, the collection of these variables may provide important information about the antithrombotic management, including the reason, the rate and the timing of crossover for each treatment.

Finally, given the evolution of the antithrombotic strategy in the last years, in particular in the pre and post Popular TAVI era, and knowing the therapeutic management during the first year of follow up, it's possible to define the impact of any study/trial on the real-world approach in recent years.

ELIGIBILITY:
Inclusion criteria

* All patients with severe aortic stenosis undergoing TAVR.
* Availability of changes in antithrombotic therapy at 1 month, 90 days, and 1 year after TAVR.

Exclusion Criteria

* Patients who died during the index procedure
* Patients in triple antithrombotic therapy at discharge
* Patients with a known prognosis less than 1 year at the time of TAVR

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with severe aortic stenosis diagnosed according to ESC guidelines, undergoing TAVR
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Trend of average daily ischemic risk (ADIR) and average daily bleeding risk (ADBR) | At 30-days, 90-days and 1 year
  ADIR was calculated as the total number of ischemic events (CV deaths, MI, ischemic stroke and other thrombotic events-including repeat events) divided by the number of patients-day at risk.
  ADBR was calculated as the total number of bleeding events (including repeat events) divided by the number of the number of patients-day at risk.
Average daily risks (ADRs) in different type of valve prosthesis | At 30-days, 90-days and 1 year
  Trend and prevalence of ADIR and ADBR in different type and number of prosthesis (long frame vs short frame, balloon versus self-expandable, porcine vs bovine, Single Valve vs Valve in Valve) and calculated as the total number of events divided by the number of patients-day at risk

SECONDARY OUTCOMES:
Average daily risks (ADRs) in different type of valve prosthesis | At 30-days, 90-days and 1 year
  Trend and prevalence of ADIR and ADBR in different type and number of prosthesis (long frame vs short frame, balloon versus self-expandable, porcine vs bovine, Single Valve vs Valve in Valve) and calculated as the total number of events divided by the number of patients-day at risk
Average daily risks (ADRs) in anaemic and thrombocytopenic patients | In hospital up to 1 year
  Trend and prevalence of ADIR and ADBR in patients who developed anaemia and thrombocytopenia after the procedure and during the hospitalization. Anaemia and thrombocytopenia were defined according to the WHO and EHA guidelines. ADRs were calculated as the total number of events divided by the number of patients-day at risk
Rate of antithrombotic regimen changes after TAVR | At 30-days, 90-days and 1 year
  Percentage of antithrombotic strategy changes
Timing of antithrombotic regimen changes after TAVR | At 30-days, 90-days and 1 year
  Number of days after the procedure in which the antithrombotic strategy was changed
Type of antithrombotic regimen changes after TAVR | At 30-days, 90-days and 1 year
  Type of changes in antithrombotic strategy taking into account all interclass (antiplatelet to anticoagulant or vice versa) and intraclass drugs switches (anticoagulant - VKA to DOAC, antiplatelet - DAPT to SAPT or vice versa)

CONTACTS AND LOCATIONS:
Locations (12):
- OLV Hospital, Aalst, Belgium
- Complejo Asistencial Dr. Sótero del Río, Santiago, Chile
- Cardiocenter, 3rd Medical School, Charles University and University Hospital Kralovske Vinohrady, Prague, Czechia
- Italy (8):
  - ASST GOM Niguarda, Milan, Italia
  - Humanitas Research Hospital, Rozzano, Milano
  - IRCCS Policlinico San Donato, San Donato Milanese, Milano
  - IRCCS Ospedale Policlinico San Martino, Genova
  - Ospedale Galeazzi Sant'Ambrogio, Milan
  - San Carlo Hospital, Potenza
  - Azienda Ospedaliera Sant'Andrea, Roma
  - A.O.U. Città della Salute e della Scienza di Torino, Torino
- Puerto Real University Hospital, Puerto Real, Cadiz, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vahanian A, Beyersdorf F, Praz F, Milojevic M, Baldus S, Bauersachs J, Capodanno D, Conradi L, De Bonis M, De Paulis R, Delgado V, Freemantle N, Gilard M, Haugaa KH, Jeppsson A, Juni P, Pierard L, Prendergast BD, Sadaba JR, Tribouilloy C, Wojakowski W; ESC/EACTS Scientific Document Group. 2021 ESC/EACTS Guidelines for the management of valvular heart disease. Eur Heart J. 2022 Feb 12;43(7):561-632. doi: 10.1093/eurheartj/ehab395. No abstract available. PMID 34453165
- [Background] Otto CM, Nishimura RA, Bonow RO, Carabello BA, Erwin JP 3rd, Gentile F, Jneid H, Krieger EV, Mack M, McLeod C, O'Gara PT, Rigolin VH, Sundt TM 3rd, Thompson A, Toly C. 2020 ACC/AHA Guideline for the Management of Patients With Valvular Heart Disease: Executive Summary: A Report of the American College of Cardiology/American Heart Association Joint Committee on Clinical Practice Guidelines. Circulation. 2021 Feb 2;143(5):e35-e71. doi: 10.1161/CIR.0000000000000932. Epub 2020 Dec 17. PMID 33332149
- [Background] Ko E, Park DW. Optimal Antithrombotic Strategy After Transcatheter Aortic Valve Replacement: Is the "Less Is More" Concept Always Better? J Am Heart Assoc. 2021 May 4;10(9):e021241. doi: 10.1161/JAHA.121.021241. Epub 2021 Apr 17. No abstract available. PMID 33870701
- [Background] Brouwer J, Nijenhuis VJ, Delewi R, Hermanides RS, Holvoet W, Dubois CLF, Frambach P, De Bruyne B, van Houwelingen GK, Van Der Heyden JAS, Tousek P, van der Kley F, Buysschaert I, Schotborgh CE, Ferdinande B, van der Harst P, Roosen J, Peper J, Thielen FWF, Veenstra L, Chan Pin Yin DRPP, Swaans MJ, Rensing BJWM, van 't Hof AWJ, Timmers L, Kelder JC, Stella PR, Baan J, Ten Berg JM. Aspirin with or without Clopidogrel after Transcatheter Aortic-Valve Implantation. N Engl J Med. 2020 Oct 8;383(15):1447-1457. doi: 10.1056/NEJMoa2017815. Epub 2020 Aug 30. PMID 32865376
- [Background] Nijenhuis VJ, Brouwer J, Delewi R, Hermanides RS, Holvoet W, Dubois CLF, Frambach P, De Bruyne B, van Houwelingen GK, Van Der Heyden JAS, Tousek P, van der Kley F, Buysschaert I, Schotborgh CE, Ferdinande B, van der Harst P, Roosen J, Peper J, Thielen FWF, Veenstra L, Chan Pin Yin DRPP, Swaans MJ, Rensing BJWM, van 't Hof AWJ, Timmers L, Kelder JC, Stella PR, Baan J, Ten Berg JM. Anticoagulation with or without Clopidogrel after Transcatheter Aortic-Valve Implantation. N Engl J Med. 2020 Apr 30;382(18):1696-1707. doi: 10.1056/NEJMoa1915152. Epub 2020 Mar 29. PMID 32223116
- [Background] Capodanno D, Collet JP, Dangas G, Montalescot G, Ten Berg JM, Windecker S, Angiolillo DJ. Antithrombotic Therapy After Transcatheter Aortic Valve Replacement. JACC Cardiovasc Interv. 2021 Aug 9;14(15):1688-1703. doi: 10.1016/j.jcin.2021.06.020. PMID 34353601
- [Background] Esposito G, Montalto C, Crimi G, Grippo R, Morici N, Bruschi G, Testa L, De Marco F, Soriano F, Nava S, Stefanini G, Bedogni F, Oreglia JA. Time course of ischemic and bleeding burden in consecutive patients undergoing transcatheter aortic valve replacement (FOCUS-ONE Registry). Int J Cardiol. 2023 Jun 15;381:2-7. doi: 10.1016/j.ijcard.2023.03.009. Epub 2023 Mar 8. PMID 36898584
- [Background] Mehran R, Baber U, Sharma SK, Cohen DJ, Angiolillo DJ, Briguori C, Cha JY, Collier T, Dangas G, Dudek D, Dzavik V, Escaned J, Gil R, Gurbel P, Hamm CW, Henry T, Huber K, Kastrati A, Kaul U, Kornowski R, Krucoff M, Kunadian V, Marx SO, Mehta SR, Moliterno D, Ohman EM, Oldroyd K, Sardella G, Sartori S, Shlofmitz R, Steg PG, Weisz G, Witzenbichler B, Han YL, Pocock S, Gibson CM. Ticagrelor with or without Aspirin in High-Risk Patients after PCI. N Engl J Med. 2019 Nov 21;381(21):2032-2042. doi: 10.1056/NEJMoa1908419. Epub 2019 Sep 26. PMID 31556978
- [Background] Valgimigli M, Frigoli E, Heg D, Tijssen J, Juni P, Vranckx P, Ozaki Y, Morice MC, Chevalier B, Onuma Y, Windecker S, Tonino PAL, Roffi M, Lesiak M, Mahfoud F, Bartunek J, Hildick-Smith D, Colombo A, Stankovic G, Iniguez A, Schultz C, Kornowski R, Ong PJL, Alasnag M, Rodriguez AE, Moschovitis A, Laanmets P, Donahue M, Leonardi S, Smits PC; MASTER DAPT Investigators. Dual Antiplatelet Therapy after PCI in Patients at High Bleeding Risk. N Engl J Med. 2021 Oct 28;385(18):1643-1655. doi: 10.1056/NEJMoa2108749. Epub 2021 Aug 28. PMID 34449185
- [Background] De Larochelliere H, Puri R, Eikelboom JW, Rodes-Cabau J. Blood Disorders in Patients Undergoing Transcatheter Aortic Valve Replacement: A Review. JACC Cardiovasc Interv. 2019 Jan 14;12(1):1-11. doi: 10.1016/j.jcin.2018.09.041. PMID 30621965